CLINICAL TRIAL: NCT04170803
Title: Feasibility of Near-infrared Spectroscopy to Measure Cortical Pain Pathway (Brain) Activation During Dry Needling
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Army-Baylor University Doctoral Program in Physical Therapy (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2018.057d; 40037-0010-0001-0208 (Other: The Geneva Foundation)
Record Dates: First submitted 2019-01-09; First posted 2019-11-20 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Shoulder Pain; Chronic Pain; Musculoskeletal Injury
Keywords: Chronic Pain; Musculoskeletal Injury; Functional near-infrared spectroscopy; Structural health monitoring; Dry needling
MeSH Terms: conditions — Shoulder Pain; Chronic Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: This study will be a randomized controlled trial. A convenience sample will be recruited from the Army Medical Department Center and School and the Brooke Army Medical Center (BAMC) Outpatient Physical Therapy Clinic using fliers and word of mouth. A computer-generated table of random numbers will be used to accomplish the group assignment. Thirty participants with shoulder pain will be randomized to receive either true or sham dry needling (Aim #1). An additional 15 participants will be recruited to receive true dry needling (Aim #2). Pre- and post-treatment and 1-week follow-up measurements will be recorded using the MyotonPRO and NIRS, in addition to measures of local hypoalgesia and self-reported pain and disability.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True Dry Needling (Experimental): Active duty DoD beneficiaries, with shoulder pain will be recruited from Army Medical Department Center and School (AMEDDC&S) and the Brooke Army Medical Center (BAMC) Outpatient Physical Therapy Clinic who meet inclusion and exclusion criteria. The TDN treatment will consist of a trained investigator inserting a needle through the participant's skin, into the infraspinatus muscle using FDA approved (FDA regulation # 880.5580) disposable 0.25 x 40 mm stainless steel Seirin J-type needles (Seirin, Japan). Each shoulder will undergo this treatment. Each needle insertion will last approximately 2-3 seconds using the "sparrow pecking" (in and out) technique to the depth of the scapula at 3 locations in the infraspinatus muscle on the affected (painful) side. When detectable, the needle insertion will specifically target palpably painful and/or "taut" bands of tissue. Immediately after use, all needles will be disposed of in approved sharps containers.
  Interventions: Device: Dry Needling
- Sham Dry Needling (Sham Comparator): The sham dry-needling procedure will mimic the dry needling procedures by placing a blunted instrument in a needling guide tube against the skin. The sharp object will be rocked and twisted to simulate treatment, but will not pierce the skin. We have used this sham dry-needling technique in previous studies performed at AMEDDC&S and have found it to be indistinguishable from real dry needling by the great majority of participants..
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Device: Dry Needling — The participant will undergo true or sham dry needling treatment with simultaneous monitoring using the NIRS head cap.
  Other Names: Trigger point dry needling; functional dry needling
  Arms: True Dry Needling
Other: Sham Dry Needling — The participant randomized to the "sham" group will undergo placebo dry needling which is functionally mimicking trigger point dry needling
  Other Names: Placebo Treatment
  Arms: Sham Dry Needling

SUMMARY:
The benefit experienced by some patients when treated with dry needling,1 combined with the field-expedient nature of this intervention, make dry needling uniquely suited for the military healthcare environment. An improved understanding of the mechanism by which dry needling exerts its clinical benefits will allow clinicians to adopt more efficacious treatment strategies for Soldiers with chronic musculoskeletal pain. The proposed study will utilize functional near-infrared spectroscopy and structural health monitoring (SHM) to provide insight on the central and peripheral mechanisms of dry needling. Phase 1 will compare the cortical pain pathway response of thirty participants with non-traumatic shoulder pain receiving either true or sham dry needling. An additional 15 participants will be enrolled to receive true dry needling to determine if brain responses may be able to predict clinical improvement (responders versus non-responders) in phase 2. Since chronic pain after musculoskeletal injury is the leading cause of medical discharge from service and a primary source of disability in the U.S. military2,3, improved complementary and alternative treatment strategies have the potential to have a large impact on both military readiness and health care costs within the Armed Forces.

DETAILED DESCRIPTION:
This study supports a line of ongoing investigation aimed at improving the diagnosis, management, and treatment of chronic pain after musculoskeletal injury. Continued progress in this arena requires novel methods to measure central nervous system (brain) mechanism of action and its role in identification of the unique transition of musculoskeletal injury to chronic pain. The purpose of this study is to use near-infrared spectroscopy (NIRS) to measure changes along cortical pain pathways in the brain related to true and sham dry needling treatment.

Specific Aim #1: The investigators will compare the cortical pain pathway response during dry needling treatment to sham dry needling treatment using NIRS in two groups of patients with chronic shoulder pain.

The investigators hypothesize that decreased cortical activity will be seen in the dorsolateral prefrontal cortex (DLPFC) in those treated with true dry needling compared to those treated with sham dry needling.

Specific Aim #2: The investigators will evaluate whether the cortical pain pathway response (imaged using NIRS) during dry needling predicts 1-week improvement in shoulder muscle response, local hypoalgesia, and self-reported pain and disability in the group of patients that received true dry needling treatment. The investigators hypothesize that decreased cortical activity in the DLPFC will be associated with improvements in shoulder muscle response, local hypoalgesia, and self-reported pain and disability in those treated with true dry needling.

ELIGIBILITY:
Inclusion Criteria:

(all of the following) Active duty DoD beneficiary Age 18-50 years old Non-traumatic shoulder pain rated at least 4/10 on the Numeric Pain Rating Scale Right-handed

Exclusion Criteria:

* Anticoagulant medication use Bleeding disorders Shoulder pain referred from cervical spine Full-thickness rotator cuff tears Known pregnancy Inability to lie prone Left- or mixed-handed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Change in Functional Near-Infrared Spectroscopy | Pre-, During intervention (real-time for approximately 3-5 minutes), directly after intervention, 1 week after intervention
  NIRS is a technology that uses low levels (less than 4mW/mm2 at 800nm) of non-ionizing, near-infrared, diffuse light to measure spectroscopic absorption changes. It will be used to non-invasively measures hemodynamic changes in the brain. An 8-channel NIRS instrument will be used to measure changes in the intensity of visible red to near-infrared light (760 and 850 nm) between sources and detectors that are placed on the scalp. Changes in intensity will be converted to optical density (absorption) and then the modified Beer-Lambert law will be applied to convert the data from optical density to change in oxy- and deoxyhemoglobin concentration.
Change in Muscle Stiffness using the MyotonPro | Pre-, directly after intervention, and 1 week after intervention
  the MyotonPRO, a research only device, (Myoton AS, Tallinn, Estonia) by applying a mechanical impulse to the skin, which is transmitted to the underlying soft tissue and muscle (0.58 N for 15 ms). 33 The oscillation of the muscle is recorded by an accelerometer located at the probe end. Measures will be taken at the same three locations in each infraspinatus muscle as the dry needling.

SECONDARY OUTCOMES:
Movement test | Pre-, directly after intervention, and 1 week after intervention
  The Hawkins-Kennedy Test - shoulder flexion and internal rotation
Change in Pain Pressure Threshold | Pre-, directly after intervention, and 1 week after intervention
  is the minimal amount of pressure that produces pain and is used to assess abnormalities in nociceptive processing or hyperalgisia.34 We will use a digital pressure algometer (Wagner Force 25 FDX, Wagner Instruments, Greenwich, CT) to measure PPT, and will operationally define it as the minimal amount of pressure that produces pain or discomfort. Pressure algometry has been found to be highly reliable, especially when using the same rater (ICC=0.94-.097)
The Global Rate of Change Score | directly after intervention and 1 week after intervention
  The GRC assesses subjective perception of overall change on a 15-point Likert type scale ranging from 1 (very great deal worse) to 15 (a very great deal better).38
Change in Numerical Pain Rating Scale | Pre-, directly after intervention, and 1 week after intervention
  will also be used to quantify clinical changes in pain. Pain during a comparable sign39 will be additionally assessed at baseline, immediately after needling, and during the follow up visit. Participants will report a simple physical maneuver that could reproduce their primary shoulder symptoms, such as shoulder flexion with internal rotation or the Hawkins-Kennedy test. Participants will then be asked to perform this maneuver and report their pain intensity using an 11-point NPRS from 0 to 10. Previous work has reported the MCID of the NPRS in patients with shoulder pain to be 1.1 points.
Pain and Shoulder Disability - The Penn Shoulder Score | Pre-,directly after intervention, and 1 week after intervention
  : The Penn Shoulder Score will be used as the primary measure of clinical outcome. This 100-point shoulder-specific self-report questionnaire consists of 3 subscales of pain, satisfaction, and function. A maximum score of 100 indicates no disability, no pain, and high satisfaction with the function of the shoulder. When aggregated, the questionnaire has demonstrated high test-retest reliability (ICC=0.94), internally consistency (Cronbach alpha = 0.93), and responsiveness in patients with shoulder pain. The minimal clinically important difference (MCID) for improvement has been reported at 11.4 points.37

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Department Center and Schools, Ft Sam Houston, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lincoln AE, Smith GS, Amoroso PJ, Bell NS. The natural history and risk factors of musculoskeletal conditions resulting in disability among US Army personnel. Work. 2002;18(2):99-113. PMID 12441574
- [Background] Koppenhaver SL, Walker MJ, Smith RW, Booker JM, Walkup ID, Su J, Hebert JJ, Flynn T. Baseline Examination Factors Associated With Clinical Improvement After Dry Needling in Individuals With Low Back Pain. J Orthop Sports Phys Ther. 2015 Aug;45(8):604-12. doi: 10.2519/jospt.2015.5801. Epub 2015 Jun 25. PMID 26110549
- [Background] Songer TJ, LaPorte RE. Disabilities due to injury in the military. Am J Prev Med. 2000 Apr;18(3 Suppl):33-40. doi: 10.1016/s0749-3797(00)00107-0. PMID 10736539
- [Background] Belmont PJ Jr, Goodman GP, Waterman B, DeZee K, Burks R, Owens BD. Disease and nonbattle injuries sustained by a U.S. Army Brigade Combat Team during Operation Iraqi Freedom. Mil Med. 2010 Jul;175(7):469-76. doi: 10.7205/milmed-d-10-00041. PMID 20684449
- [Background] Galanter M, Dermatis H, Sampson C. Narcotics anonymous: a comparison of military veterans and non-veterans. J Addict Dis. 2014;33(3):187-95. doi: 10.1080/10550887.2014.950031. PMID 25115224
- [Background] Vanderlip ER, Sullivan MD, Edlund MJ, Martin BC, Fortney J, Austen M, Williams JS, Hudson T. National study of discontinuation of long-term opioid therapy among veterans. Pain. 2014 Dec;155(12):2673-2679. doi: 10.1016/j.pain.2014.09.034. Epub 2014 Sep 30. PMID 25277462
- [Background] Mosher HJ, Krebs EE, Carrel M, Kaboli PJ, Weg MW, Lund BC. Trends in prevalent and incident opioid receipt: an observational study in Veterans Health Administration 2004-2012. J Gen Intern Med. 2015 May;30(5):597-604. doi: 10.1007/s11606-014-3143-z. Epub 2014 Dec 18. PMID 25519224
- [Background] Jonas WB, Schoomaker EB. Pain and opioids in the military: we must do better. JAMA Intern Med. 2014 Aug;174(8):1402-3. doi: 10.1001/jamainternmed.2014.2114. No abstract available. PMID 24978149
- [Background] Petri RP Jr. Integrative Health and Healing as the New Health Care Paradigm for the Military. Med Acupunct. 2015 Oct 1;27(5):301-308. doi: 10.1089/acu.2014.1068. PMID 26543516
- [Background] Thomas DA, Maslin B, Legler A, Springer E, Asgerally A, Vadivelu N. Role of Alternative Therapies for Chronic Pain Syndromes. Curr Pain Headache Rep. 2016 May;20(5):29. doi: 10.1007/s11916-016-0562-z. PMID 27038968
- [Background] Clarke TC, Black LI, Stussman BJ, Barnes PM, Nahin RL. Trends in the use of complementary health approaches among adults: United States, 2002-2012. Natl Health Stat Report. 2015 Feb 10;(79):1-16. PMID 25671660
- [Background] Sherman KJ, Cherkin DC, Eisenberg DM, Erro J, Hrbek A, Deyo RA. The practice of acupuncture: who are the providers and what do they do? Ann Fam Med. 2005 Mar-Apr;3(2):151-8. doi: 10.1370/afm.248. PMID 15798042
- [Background] Cummings TM, White AR. Needling therapies in the management of myofascial trigger point pain: a systematic review. Arch Phys Med Rehabil. 2001 Jul;82(7):986-92. doi: 10.1053/apmr.2001.24023. PMID 11441390
- [Background] Boyles R, Fowler R, Ramsey D, Burrows E. Effectiveness of trigger point dry needling for multiple body regions: a systematic review. J Man Manip Ther. 2015 Dec;23(5):276-93. doi: 10.1179/2042618615Y.0000000014. PMID 26955257
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] Zhou K, Ma Y, Brogan MS. Dry needling versus acupuncture: the ongoing debate. Acupunct Med. 2015 Dec;33(6):485-90. doi: 10.1136/acupmed-2015-010911. Epub 2015 Nov 6. PMID 26546163
- [Background] Vulfsons S, Ratmansky M, Kalichman L. Trigger point needling: techniques and outcome. Curr Pain Headache Rep. 2012 Oct;16(5):407-12. doi: 10.1007/s11916-012-0279-6. PMID 22610507
- [Background] Hsieh YL, Chou LW, Joe YS, Hong CZ. Spinal cord mechanism involving the remote effects of dry needling on the irritability of myofascial trigger spots in rabbit skeletal muscle. Arch Phys Med Rehabil. 2011 Jul;92(7):1098-105. doi: 10.1016/j.apmr.2010.11.018. Epub 2011 May 6. PMID 21529778
- [Background] Koppenhaver SL, Walker MJ, Su J, McGowen JM, Umlauf L, Harris KD, Ross MD. Changes in lumbar multifidus muscle function and nociceptive sensitivity in low back pain patient responders versus non-responders after dry needling treatment. Man Ther. 2015 Dec;20(6):769-76. doi: 10.1016/j.math.2015.03.003. Epub 2015 Mar 13. PMID 25801100
- [Background] Cagnie B, Barbe T, De Ridder E, Van Oosterwijck J, Cools A, Danneels L. The influence of dry needling of the trapezius muscle on muscle blood flow and oxygenation. J Manipulative Physiol Ther. 2012 Nov-Dec;35(9):685-91. doi: 10.1016/j.jmpt.2012.10.005. PMID 23206963
- [Background] Aird L, Samuel D, Stokes M. Quadriceps muscle tone, elasticity and stiffness in older males: reliability and symmetry using the MyotonPRO. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):e31-9. doi: 10.1016/j.archger.2012.03.005. Epub 2012 Apr 13. PMID 22503549
- [Background] Ylinen J. Pressure algometry. Aust J Physiother. 2007;53(3):207. doi: 10.1016/s0004-9514(07)70032-6. No abstract available. PMID 17899675
- [Background] Leggin BG, Michener LA, Shaffer MA, Brenneman SK, Iannotti JP, Williams GR Jr. The Penn shoulder score: reliability and validity. J Orthop Sports Phys Ther. 2006 Mar;36(3):138-51. doi: 10.2519/jospt.2006.36.3.138. PMID 16596890
- [Background] Takamoto K, Hori E, Urakawa S, Sakai S, Ishikawa A, Kohno S, Ono T, Nishijo H. Cerebral hemodynamic responses induced by specific acupuncture sensations during needling at trigger points: a near-infrared spectroscopic study. Brain Topogr. 2010 Sep;23(3):279-91. doi: 10.1007/s10548-010-0148-8. Epub 2010 May 26. PMID 20502956
- [Background] Huppert TJ. Commentary on the statistical properties of noise and its implication on general linear models in functional near-infrared spectroscopy. Neurophotonics. 2016 Jan;3(1):010401. doi: 10.1117/1.NPh.3.1.010401. Epub 2016 Mar 2. PMID 26989756